CLINICAL TRIAL: NCT07391423
Title: Assessing Psoriasis Treatment Outcomes: a Single-center, Prospective Study Evaluating Patient Outcomes in Psoriasis
Brief Title: Assessing Psoriasis Treatment Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00142799
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: Psoriasis Treatment Outcomes; medication adherence; Artificial intelligence
MeSH Terms: conditions — Psoriasis; Medication Adherence | interventions — Artificial Intelligence; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI intervention group (Experimental): Subject will receive with topical betamethasone dipropionate cream (BD) and have a weekly virtual visit with an AI-generated automated physician provider (AIGPP).
  Interventions: Behavioral: Artificial intelligence
- Human intervention group (Experimental): Subjects will receive BD and receive weekly video calls from study staff
  Interventions: Behavioral: Human
- Standard of Care Group (Other): Subjects will receive BD and scheduled for a single follow up visit in 4 weeks
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Artificial intelligence — patients will receive BD and have a weekly virtual visit with an AIGPP
  Other Names: Artificial intelligence (AI)
  Arms: AI intervention group
Behavioral: Human — patients will receive BD and receive weekly video calls from study staff
  Arms: Human intervention group
Other: Standard of Care — patients will receive BD and scheduled for a single follow up visit in 4 weeks
  Arms: Standard of Care Group

SUMMARY:
To assess the feasibility of AIGPP video interactions with psoriasis patients. To explore patient attitudes, trust, and comfort levels concerning AIGPP interactions in a healthcare setting, and to understand their influence on the patient-physician dynamic. To evaluate medication adherence over a 4-week period in patients with psoriasis randomized to weekly AI-generated automated physician providers (AIGPP) video interactions, weekly human video calls, or standard care (single follow up visit after 4 weeks). Adherence rates will be evaluated via a cap designed to record adherence attached to the study medication container.

DETAILED DESCRIPTION:
Psoriasis is a chronic disease that can negatively impact quality of life. However, adherence to topical treatment for psoriasis can be abysmal. Nonadherence can result in multiple negative effects, including treatment failure, increased healthcare costs, and decreased quality of life. Office visits can drive compliance behavior. By using "white coat compliance," providers increase adherence in the short period before and after a doctor appointment. However, frequent visits may not be feasible for time-constrained healthcare providers. Artificial intelligence (AI) has alleviated provider burden in other settings and may be applied in promoting medication adherence through AI-generated automated physician provider (AIGPP) visits. Given limited funding, this pilot study will assess the feasibility of AIGPP interactions with psoriasis patients treated with betamethasone dipropionate cream (BD).

To accomplish this, up to 15 subjects, age 18 years of age and older, with psoriasis will be recruited to participate. Subjects who meet inclusion criteria will complete a demographic questionnaire and will be randomized to one of three arms (1. AI intervention group - patients will receive BD and have a weekly virtual visit with an AIGPP, 2. human intervention group - patients will receive BD and receive weekly video calls from study staff, 3. standard of care group - patients will receive BD and scheduled for a single follow up visit in 4 weeks). The subjects will receive the BD with a Sensal MyAide adherence device attached.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Patients with a current diagnosis of psoriasis suitable for treatment with topical Betamethasone (BD)
* Patients who live in the United States
* Patients with a sufficient command of the English language
* Patients with a mobile device able to at least operate at 25 frames per second (FPS).

Exclusion Criteria:

* Patients less than the age of 18
* Patients with severe or unstable comorbid conditions
* Patient who are pregnant or breastfeeding
* Patients with any other skin conditions that prohibit or confound the ability of the investigator to interpret skin findings
* Patients that are taking concomitant topical or systemic therapy for the treatment of psoriasis and/or phototherapy
* Patients without mobile devices able to at least operate at 25 frames per second (FPS).
* Patients without a current diagnosis of psoriasis suitable for treatment with topical BD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Ability to implement AIGPP system and Rate of dropout in AIGPP trial arm | Week 4
  One primary outcome of the study is the feasibility of AIGPP interactions with psoriasis patients, which will be measured as whether we can create & implement the AIGPP system and the dropout rate in the AIGPP arm
Thematic analysis of qualitative interviews regarding psoriasis patients' attitudes, trust, and comfort levels with AIGPP interactions in a healthcare setting | Week 4
  Another primary outcome will be psoriasis patients' attitudes, trust, and comfort levels with AIGPP interactions in a healthcare setting, which will be measured by semi-structured qualitative interviews analyzed via a thematic analysis.

SECONDARY OUTCOMES:
Rate of Adherence | Week 4
  One secondary outcome is adherence, which will be measured as a continuous variable as the number of days the study medication is used divided by the number of study days.
Rate of PASI75, PASI90, PASI100, and IGA of 0 or 1 | Baseline, Week 4
  Another secondary outcome is efficacy, which will be measured as 75% improvement in Psoriasis Area and Severity Index (PASI75), 90% improvement in PASI (PASI90), and 100% improvement in PASI (PASI100). Efficacy will also be measured as the rate of Investigator Global Assessment (IGA) of 0 (clear) and 1 (almost clear)
Rate of adverse events | Week 4
  Another secondary outcome will be adverse events, which will be assessed at the study conclusion and will be patient reported.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, M.D., Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No